CLINICAL TRIAL: NCT06640413
Title: A Phase I Study to Evaluate the Safety and Preliminary Signs of Efficacy of [177Lu]Lu-OncoFAP-23 Alone or in Combination With L19-IL2 as a Treatment of Metastatic FAP-positive Solid Tumors
Brief Title: A Study to Evaluate the Safety and Preliminary Signs of Efficacy of [177Lu]Lu-OncoFAP-23 Alone or in Combination With L19-IL2 as a Treatment of Metastatic FAP-positive Solid Tumors
Acronym: TheraTri
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-FAPLU-02/23; 2023-509453-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: FAP
Keywords: Patients with advanced/metastatic FAP-positive tumors

STUDY DESIGN:
Intervention Model Description: In Part I patients are assigned to 5 sequential dose escalation cohorts. In this part, two arms are foreseen:
  Arm 1 foresees cohort 1-3 with monotherapy of [177Lu]Lu-OncoFAP-23 (3.7, 7.4, 11.1 GBq respectively); Arm 2, only opened when the MTD and RD is established, has cohorts 4-5 that are run with [177Lu]Lu-OncoFAP-23 in combination with L19IL2 at 22.5 Mio International Units (IU).
  In Part II, 10 patients are randomly assigned to Arm 1 (monotherapy of [177Lu]Lu-OncoFAP-23 at the recommended dose) and 10 patients are randomly assigned to Arm 2 (combination of [177Lu]Lu-OncoFAP-23 and L19IL2 at the recommended doses).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Part I - Dose Escalation - Cohort 1, Arm 1 (Experimental): In Arm 1, patients assigned to this cohort 1, receive monotherapy of [177Lu]Lu-OncoFAP-23 (3.7 GBq)
  Interventions: Drug: [177Lu]Lu-OncoFAP-23
- Part I - Dose Escalation - Cohort 2, Arm 1 (Experimental): In Arm 1, patients assigned to this cohort 2, receive monotherapy of [177Lu]Lu-OncoFAP-23 (7.4 GBq)
  Interventions: Drug: [177Lu]Lu-OncoFAP-23
- Part I - Dose Escalation - Cohort 3, Arm 1 (Experimental): In Arm 1, patients assigned to this cohort 3, receive monotherapy of [177Lu]Lu-OncoFAP-23 (11.1 GBq)
  Interventions: Drug: [177Lu]Lu-OncoFAP-23
- Part I - Dose Escalation - Cohort 4, Arm 2 (Experimental): In Arm 2, patients assigned to this cohort 4, receive combination of [177Lu]Lu-OncoFAP-23 at at the dose level below the Maximum Tolerated Dose (MTD) with L19IL2 (22.5 Mio IU).
  Interventions: Drug: [177Lu]Lu-OncoFAP-23; Drug: L19IL2
- Part I - Dose Escalation - Cohort 5, Arm 2 (Experimental): In Arm 2, patients assigned to this cohort 4, receive combination of [177Lu]Lu-OncoFAP-23 at MTD with L19IL2 (22.5 Mio IU).
  Interventions: Drug: [177Lu]Lu-OncoFAP-23; Drug: L19IL2
- Part II - Dose Expansion - Arm 1 (Experimental): 10 patients receive the monotherapy of [177Lu]Lu-OncoFAP-23 at the recommended dose
  Interventions: Drug: [177Lu]Lu-OncoFAP-23
- Part II - Dose Expansion - Arm 2 (Experimental): 10 patients receive the combination of [177Lu]Lu-OncoFAP-23 and L19IL2 at the recommended doses
  Interventions: Drug: [177Lu]Lu-OncoFAP-23; Drug: L19IL2

INTERVENTIONS:
Drug: [177Lu]Lu-OncoFAP-23 — 3.7, 7.4, or 11.1 GBq to define the RD
Drug: L19IL2 — 22.5 Mio IU
  Arms: Part I - Dose Escalation - Cohort 4, Arm 2; Part I - Dose Escalation - Cohort 5, Arm 2; Part II - Dose Expansion - Arm 2

SUMMARY:
The aim of this study is to assess the safety of [177Lu]Lu-OncoFAP-23 alone or in combination with L19-IL2 for the treatment of advanced/metastatic Fibroblast Activation Protein (FAP)-positive solid tumors and to establish a Recommended Dose (RD).

DETAILED DESCRIPTION:
This study is a prospective phase I, open-label, multiple ascending, multi-center dose escalation study to evaluate the safety and preliminary signs of efficacy of [177Lu]Lu-OncoFAP-23 alone and in combination with the antibody-cytokine conjugate L19-IL2 for the treatment of advanced/metastatic FAP-positive solid tumors.

Eligible patients for this trial are male or non-pregnant and non-breastfeeding females aged 18 years or more, able to give informed consent.

Up to 56 evaluable patients will be enrolled in the trial and the trial is divided into two parts:

1. Part I - Dose escalation part (2-36 pts) This dose escalation part of the study is designed as a standard 3+3 escalation scheme. Not more than 2 patients per cohort are treated simultaneously during the Dose Limiting Toxicity (DLT) observation period from Day 1 to Day 28 of the first cycle. Patients per cohort will be assigned to different dose levels of the study drug.
2. Part II - Dose expansion part (20 pts) After completion of the dose escalation part, additional 20 patients will be enrolled at the RD to better understand the safety profile and to explore early signs of efficacy in different disease indications. Patients will be randomly assigned to arm 1 (monotherapy) or arm 2 (combination therapy) (10 patients each).

Both in part I and II, patients can receive up to 4 consecutive cycles of radioligand therapy every 8 (± 1) weeks.

The primary objective of this study is to assess the safety of [177Lu]Lu-OncoFAP-23 alone or in combination with L19-IL2 for the treatment of advanced/metastatic FAP-positive malignancies and to establish a Recommended Dose (RD).

Secondary objectives include evaluation of pharmacokinetics and the collection of initial signs of efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced/metastatic solid tumors, who have progressed on available standard treatments.
2. Patients with FAP-positive tumors as evaluated by [68Ga]Ga-OncoFAP-DOTAGA-PET/CT imaging.
3. Patients without other therapeutic alternatives with curative or survival prolonging potential as per investigator judgement.
4. Male or non-pregnant and non-breast feeding female, age 18 or more.
5. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria 1.1. This lesion should not have been irradiated during previous treatments.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
7. Survival expectation of more than 12 weeks.
8. Ability to undergo standard imaging.
9. Documented negative test for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV). For HBV serology: the determination of HBsAg and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBsAg-Ab with no history of vaccination and/or anti-HBcAg-Ab), negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
10. All acute toxic effects (excluding alopecia and fatigue) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v. 5.0) Grade ≤ 1.
11. Female patients: negative blood pregnancy test at Screening for women of childbearing potential (WOCBP)*. WOCBP must agree to use, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the Recommendations for contraception and pregnancy testing in clinical ; issued by the Head of Medicine Agencies; Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.
12. Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g., condom with spermicidal gel). Double-barrier contraception is required.
13. A personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and has given consent to participate in the study.
14. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

1. Any cancer therapy within 4 weeks of study entry.
2. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent.
3. Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, Iodine-131, Lutetium-177 conjugates or hemi-body irradiation within 6 months prior to enrollment.
4. White blood cell count (WBC) minor than 2.5 x 109/L, absolute neutrophil count (ANC) minor than 1.5 x 109/L, platelets minor than 100 x 109/L or hemoglobin (Hb) minor than 9.0 g/dl,
5. Chronically impaired renal function as expressed by creatinine clearance minor than 60 mL/min or serum creatinine major than 1.5 ULN.
6. Inadequate liver function (Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 3 x Upper Limit of Normal (ULN), or Alkaline Phosphatase (ALP) or Gamma Glutamyl Transferase (GGT) ≥ 2.5 x ULN, or total bilirubin ≥ 1.5 x ULN). For patients with metastatic lesions in the liver ALT, AST, GGT or ALP ≥ 5 x ULN.
7. Presence of cirrhosis or active hepatitis.
8. Patients with Central Nervous System (CNS) metastases.
9. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
10. Heart insufficiency (major Grade II, New York Heart Association (NYHA) criteria).
11. Clinically significant cardiac arrhythmias or requiring permanent medication.
12. Abnormal Left Ventricular Ejection Fraction (LVEF) or any other abnormalities observed during baseline Electrocardiogram (ECG) and echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current, or a history of QT/QTc prolongation would be excluded. In particular: - patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc major than 480 milliseconds using Fredricia's QT correction formula) are excluded; - patients with a history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of prolonged QT syndrome) are excluded; - patients who require the use of concomitant medications that prolong the QT/QTc interval are excluded.
13. Cardioversion in the previous 12 months
14. Uncontrolled hypertension as defined by systolic blood pressure ≥ 140 mmHg and diastolic blood pressure ≥ 90 mmHg at 3 consecutive measurements performed within one week. Note: if the first blood pressure measurement is below threshold for systolic or diastolic blood pressure, it is not required to repeat the measurement.
15. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
16. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
17. Pregnancy or lactation or unwillingness to use adequate method of birth control.
18. Any severe concomitant condition which in the opinion of investigators makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
19. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of the study drug.
20. Serious, non-healing wound, ulcer or bone fracture.
21. Known history of allergy to an excipient in study medication or any other intravenously administered human proteins/peptides/antibodies
22. Systemic chronic steroid therapy (major than 10 mg/day prednisone or equivalent) or any other immunosuppressive therapy within 14 days prior to study treatment start. Topical, inhaled, nasal and ophthalmic steroids are allowed.
23. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
24. Concurrent or previous malignancies (other than the indication for this trial), unless a complete remission without further recurrence was achieved at least 2 years prior to study treatment start.
25. Growth factors or immunomodulatory agents within 7 days prior to study treatment start.
26. Deep vein thrombosis, pulmonary embolism, or other acute vascular events within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | From Day 1 to 28 of the dose escalation part
  Dose Limiting Toxicity (DLT)
Maximum Tolerated Dose (MTD) and Recommended Dose (RD) | From Day 1 to 28 of the dose escalation part
  Maximum Tolerated Dose (MTD) and Recommended Dose (RD)
Maximum Administered Dose (MAD) | From Day 1 to 28 of the dose escalation part
  Maximum Administered Dose (MAD)
Adverse Events (AEs) and Serious Adverse Events (SAEs) | through study completion, maximum 1 year
  Adverse events (AEs) and Serious Adverse Events (SAEs) assessment based on Common Terminology Criteria for Adverse Events v. 5.0 (CTCAE)
Drug Induced Liver Injury (DILI) | through study completion, maximum 1 year
  Drug Induced Liver Injury (DILI) assessment based on Common Terminology Criteria for Adverse Events v. 5.0 (CTCAE)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - ASST Papa Giovanni XXIII Piazza OMS, Bergamo, Bergamo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano
  - Istituto Europeo di Oncologia, Milan, Milano
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale" Via Mariano Semmola, Napoli, Napoli

IPD SHARING:
Plan to Share IPD: No